CLINICAL TRIAL: NCT06302725
Title: Vaginal Self-sampling for Detecting High-risk Human Papillomavirus Cervical Infection in Patients With Immune-mediated Inflammatory Diseases
Acronym: APOSY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: APHP231514; 2023-A02623-42 (Other: IDRCB)
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: HPV Infection; Systemic Disease
Keywords: HPV; systemic disease; cervical cancer screening; vaginal self sampling
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vaginal self sampling detecting HPV (Experimental)
  Interventions: Procedure: Vaginal self sampling detecting HPV

INTERVENTIONS:
Procedure: Vaginal self sampling detecting HPV — IMIDs patients who are not up to date with CCS be included into the study to perform a vaginal self-screening (VSS) A positive VSS will be confirmed by a standard HPV test and management of the results of standard HPV test or VSS will be performed as planned following HAS guidelines. For women with a positive VSS, follow-up results (HPV test and cytology, biopsy, etc.) will be collected according to the usual procedures of the screening facility and in accordance with the recommendations of the Health authorities

SUMMARY:
Main objective: -To determine Human Papilloma Virus (HPV) prevalence in patients with immune-mediated inflammatory diseases (IMID) using vaginal self-sampling (VSS), one year after VSS was proposed Primary endpoint: - To determine the prevalence of HPV infection (yes/no) after VSS proposal Secondary objectives: - To describe the HPV typology and the rate of co-infection (with several high-risk HPV (HR-HPV)) in this population - To describe the factors associated with the presence of HPV infection - To determine the rate of HPV clearance after one year, during the second screening at 12 months- To determine the percentage of pre-cancerous cervical lesions and cervical cancer in the event of subsequent cervical smear - To determine the factors associated with persistence (or non-clearance ) of HPV infection - To determine the factors associated with the presence of pre-cancerous and cancerous cervical lesions - To determine the characteristics, tolerance and acceptability of VSS - To determine the rate of cervical cancer screening carried out following French Health Authorities guidelines -To determine the HPV vaccination coverage Secondary endpoints: 1/ HPV typology and presence of co-infection (Yes/No, type) or HPV multi-infection (more than 2 HPV, Yes/No) identified on samples at inclusion and at 1 year. 2/ Explanatory variables: demographic, clinical, biological factors and treatments (corticoids, immunosuppressive treatments); variable to be explained: presence of HPV infection during follow-up. 3/ Characteristics, acceptability, obstacles and tolerance of VPA reported by self-questionnaire (including procedure failures, bleeding and pain). 4/ Up-to-date cervical cancer screening rate in accordance with HAS recommendations at 12 months post-procedure. 5/ Proportion of cervical cytological abnormalities and cervical cancer authenticated on cervico-vaginal smear, if performed (histological confirmation if available) during follow-up. 6/ Explanatory variables: demographic, clinical, biological factors and treatments (corticoids, immunosuppressants; variable to be explained: presence of cervical precancerous lesions and cervical cancer, authenticated on cervico-vaginal smear, if performed (histological confirmation if available) during follow-up. 7/ HPV vaccination coverage rate (measured on initial self-questionnaire) 8/ Prevalence of HR-HPV(s) at second screening at one year, in the case of initial positivity (Persistence of HPV infection (Yes/No). 9/ Explanatory variables: demographic, clinical, biological factors and treatments (corticoids, immunosuppressive treatments); variable to be explained: persistence of cervical HPV infection at one year (in the case of initial positivity).

ELIGIBILITY:
Inclusion Criteria:

Prospective and retrospective patient

* Women aged 30 to 65 years old
* presenting with MSIA, MSIA includes Systemic lupus erythematosus Sjögren's syndrome Systemic scleroderma Mixed connective tissue disease Inflammatory myositis Systemic sarcoidosis Systemic vasculitis Behçet's disease Adult-onset Still's disease IgG4-related disease Autoimmune cytopenia (autoimmune hemolytic anemia, immune thrombocytopenic purpura, Evans syndrome) Susac syndrome
* Followed in the internal medicine department of Bichat Hospital, Paris
* Not up to date with gynecological follow-up (i.e., Pap smear more than one year old or undatable) (for retrospective patients: at the time of initial screening)

Retrospective patient

- Patient who underwent Pap smear screening less than one year before the start of the study

Exclusion Criteria:

Prospective and retrospective patient

* Patient under legal protection, guardianship, or trusteeship
* History of colpohysterectomy
* Not affiliated with a social security scheme (general or CMU)
* Absence of informed and written consent

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
prevalence of HPV infection (yes/no) after VSS proposal | at one year

SECONDARY OUTCOMES:
the HPV typology of co-infection (with several high-risk HPV (HR-HPV)) in this population | at inclusion and at one year after inclusion
The rate of co-infection (with several high-risk HPV (HR-HPV)) in this population | at inclusion and at one year after inclusion

OTHER OUTCOMES:
Presence of HPV infection during follow-up (yes/no) | at inclusion and at one year
description of demographic factor | at inclusion and at one year
description of clinical factor | at inclusion and at one year
description of biological factor | at inclusion and at one year
description of treatment (corticoids, immunosuppressive treatments) | at inclusion and at one year
description of characteristics of VPA reported by self-questionnaire (including procedure failures, bleeding and pain). | at inclusion and at one year
description of acceptability of VPA reported by self-questionnaire (including procedure failures, bleeding and pain). | at inclusion and at one year
description of tolerance of VPA reported by self-questionnaire (including procedure failures, bleeding and pain). | at inclusion and at one year
description obstacles of VPA reported by self-questionnaire (including procedure failures, bleeding and pain). | at inclusion and at one year
Up-to-date cervical cancer screening rate in accordance with HAS recommendations | at 12 months post-inclusion.
Proportion of cervical cytological abnormalities if performed (histological confirmation if available) | during 1 year of follow-up
proportion of cervical cancer authenticated on cervico-vaginal smear, if performed (histological confirmation if available) | during 1 year of follow-up
presence of cervical precancerous lesions and cervical cancer | during 1 year of follow-up
  authenticated on cervico-vaginal smear, if performed (histological confirmation if available)
HPV vaccination coverage rate | at inclusion
  (measured on initial self-questionnaire)
Persistence of HPV infection | at one year
  Prevalence of HR-HPV(s) at second screening , in the case of initial positivity

CONTACTS AND LOCATIONS:
Overall Officials: Tiphaine Goulenok, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Service de Médecine Interne - Hôpital Bichat Claude Bernard, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Goulenok T, Sacre K. HPV Infection and Prevention in Patients With Immune-Mediated Inflammatory Diseases: A Scoping Review. J Clin Rheumatol. 2024 Oct 1;30(7S Suppl 1):S34-S41. doi: 10.1097/RHU.0000000000002122. PMID 39325123